CLINICAL TRIAL: NCT01183923
Title: Dietary Interventions in Asthma Treatment: Sprouts Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Environmental Health Sciences (NIEHS) (NIH); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NA_00035087; 1P01ES018176-01 (NIH)
Record Dates: First submitted 2010-08-17; First posted 2010-08-18 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Asthma; Allergy
Keywords: asthma; dietary interventions; mouse allergy
MeSH Terms: conditions — Asthma; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Broccoli Sprouts, then Alfalfa Sprouts (Experimental): Broccoli Sprout sandwich/wrap will be eaten daily for 7 consecutive days followed by alfalfa sprouts after washout.
  Interventions: Other: Broccoli Sprouts; Other: Alfalfa Sprouts
- Alfalfa Sprouts, then Broccoli Sprouts (Experimental): Alfalfa Sprout sandwich/wrap will be eaten daily for 7 consecutive days followed by broccoli sprouts after washout.
  Interventions: Other: Broccoli Sprouts; Other: Alfalfa Sprouts

INTERVENTIONS:
Other: Broccoli Sprouts — Broccoli Sprouts will be eaten daily in a sandwich form during the intervention period for broccoli sprouts.
Other: Alfalfa Sprouts — Alfalfa sprouts will be eaten daily in a sandwich form during the intervention period for alfalfa sprouts.

SUMMARY:
Sulforaphane (SFN) is a naturally occurring isothiocyanate that is a potent inducer of Phase II enzymes which play a critical role in preventing oxidative stress (via activation of Nrf2). Broccoli sprouts (BS) contain the richest source of SFN.

The main objectives of this study are to test the effect of broccoli sprouts (BS) on biomarkers of oxidative stress (OS), inflammation, basophil activation, and clinical outcomes in mouse allergen-induced asthma by (1) determining if BS improves lung function and airways symptom responses in mouse-sensitized adults with asthma undergoing environmental mouse allergen challenge (EMAC), (2) examining the effect of BS on OS, inflammation, and basophil activation, and (3) examining the effect of BS on changes in OS, inflammation, and basophil activation after EMAC.

DETAILED DESCRIPTION:
After eligibility is confirmed, participants will be randomized to (a) placebo then BS or (b) BS then placebo. At randomization, baseline exhaled nitric oxide (eNO), forced expiratory volume at one second (FEV1), nasal epithelial gene expression, urinary OS biomarkers, serum inflammatory and OS biomarkers, and basophil activation will be assessed. These will be assessed again after 7 days on the assigned intervention at two time points: pre- and post-EMAC. The 1 week time period was chosen because previous studies have shown that daily ingestion of a broccoli sprout homogenate for three days resulted in upregulation of phase II enzyme gene expression in nasal epithelial cells. Following a 2-week washout period, this protocol will be repeated for the second intervention, phase II. The 2 week washout period will be sufficient as the half life of the extract of the active ingredient in broccoli sprouts, SFN, has been shown to be 1.8 hours.(16) Participants' diets will be assessed before and after each intervention with a Food Frequency Questionnaire and a questionnaire to capture intake of specific foods that are rich in SFN.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-49 years
* Physician-diagnosed asthma
* No other major pulmonary disease such as cystic fibrosis or chronic obstructive pulmonary disease (COPD)
* Mouse sensitization, defined by a positive skin prick test to mouse epithelial extract or positive mouse-specific immunoglobulin E (IgE)
* Non-smoker

Exclusion Criteria:

* Severe or unstable asthma defined as requiring hospitalization in the previous year or intubation in the previous 2 years, or on high-dose inhaled corticosteroids or chronic oral corticosteroids
* Baseline FEV1 and FEV1/forced vital capacity (FVC) < 70% predicted
* Positive skin prick test (SPT) to a pet currently living in the participant's home
* Other significant medical issues such as heart disease or poorly controlled hypertension, or hypothyroidism
* Pregnancy or nursing/breastfeeding mothers
* On beta-blocker therapy
* Taking anti-oxidant supplements
* Unable to stop antihistamines prior to skin testing
* Unable to stop medications that may interfere with allergen challenge responses prior to challenges.
* The participant has food allergy to BS or AS.
* Omalizumab use within the last 12 months.
* Oral corticosteroid use within the last 2 weeks.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2010-11; Primary Completion 2012-02-06 (Actual); Study Completion 2012-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Matsui, MD MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Sudini K, Diette GB, Breysse PN, McCormack MC, Bull D, Biswal S, Zhai S, Brereton N, Peng RD, Matsui EC. A Randomized Controlled Trial of the Effect of Broccoli Sprouts on Antioxidant Gene Expression and Airway Inflammation in Asthmatics. J Allergy Clin Immunol Pract. 2016 Sep-Oct;4(5):932-40. doi: 10.1016/j.jaip.2016.03.012. Epub 2016 Apr 27. PMID 27130714

RESULTS

PARTICIPANT FLOW:
Groups:
- Broccoli Sprouts, Then Alfalfa Sprouts: Broccoli Sprouts will be eaten daily in a sandwich form, followed by a 14 day washout, and then alfalfa sprouts will be eaten daily in a sandwich form.
- Alfalfa Sprouts, Then Broccoli Sprouts: Alfalfa sprouts will be eaten daily in a sandwich form, followed by a 14 day washout, and then broccoli sprouts will be eaten daily in a sandwich form.
Period: Intervention 1 (7 Days)
Arm/Group | Broccoli Sprouts, Then Alfalfa Sprouts | Alfalfa Sprouts, Then Broccoli Sprouts
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0
Period: Washout (14 Days)
Arm/Group | Broccoli Sprouts, Then Alfalfa Sprouts | Alfalfa Sprouts, Then Broccoli Sprouts
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0
Period: Intervention 2 (7 Days)
Arm/Group | Broccoli Sprouts, Then Alfalfa Sprouts | Alfalfa Sprouts, Then Broccoli Sprouts
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: the study population will be randomized in a 1:1 ratio to first eat broccoli sprouts followed by a washout period and then eat alfalfa sprouts, or to start with alfalfa sprouts followed by a washout and then eat broccoli sprouts
Arm/Group | All Participants
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Forced Expiratory Volume at One Second (FEV1)
Description: The percentage change in FEV1 from the pre-challenge FEV1 value over the 1 hour mouse chamber exposure.
Time Frame: 30 days
Population: Trial was halted due to an adverse event after the second intervention. The participant could not complete the second challenge for data to be obtained.
Measure: Number; unit: percent change
Groups:
- Broccoli Sprouts: Broccoli Sprouts: Broccoli Sprouts will be eaten daily in a sandwich form followed by a washout period, after which alfalfa sprouts will be eaten in a sandwich form.
- Alfalfa Sprouts: Participants who received alfalfa sprouts
Arm/Group | Broccoli Sprouts | Alfalfa Sprouts
Number analyzed (Participants) | 1 | 0
percent change | -18 |

ADVERSE EVENTS:
Groups:
- Total Study Population: Total population, which is randomized 1:1 to broccoli sprouts, then alfalfa sprouts or alfalfa sprouts, then broccoli sprouts
Arm/Group | Total Study Population
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Study Population (N=1)
bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No